CLINICAL TRIAL: NCT03395678
Title: Comparison of Fractionated 1,540nm Nonablative Laser and Microneedling in the Treatment of Atrophic Acne Scarring in Skin of Color: A Randomized Controlled Study
Brief Title: Acne Scarring in Skin of Color: Laser vs Microneedling
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sample size can not be obtained at this site.
Sponsor: Boston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-37256
Record Dates: First submitted 2018-01-04; First posted 2018-01-10 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Acne Vulgaris; Scar
Keywords: Microneedling; Nonablative fractional lasers; Fitzpatrick skin types III-V; Arophic acne scarring
MeSH Terms: conditions — Acne Vulgaris; Cicatrix | interventions — Percutaneous Collagen Induction; Lasers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Microneedling (Experimental): Participants in this arm will receive 5 treatments of microneedling.
  Interventions: Device: Microneedling
- Fractional non-ablative 1,540nm laser (Active Comparator): Participants in this arm will receive 5 treatments of fractional non-ablative1,540nm laser.
  Interventions: Device: Fractional non-ablative 1,540nm laser

INTERVENTIONS:
Device: Microneedling — The exact microneedling settings will be tailored to each patient based on skin type, photodamage, skin thickness based on area of the face. Settings will be adjusted to deliver similar endpoints among all patients. Each participant will receive 5 treatments a month apart.
  Other Names: DermaPen 3MD
  Arms: Microneedling
Device: Fractional non-ablative 1,540nm laser — The exact laser settings will be tailored to each patient based on skin type, photodamage, skin thickness based on area of the face. Settings will be adjusted to deliver similar endpoints among all patients. Each participant will receive 5 treatments a month apart.
  Other Names: Palomar StarLux
  Arms: Fractional non-ablative 1,540nm laser

SUMMARY:
Atrophic acne scars are a common and important sequelae of acne that affect up to 43-55% of patients with acne. Scarring impacts quality of life with reports of diminished self-esteem and frustration/sadness; additionally, some individuals report that their appearance even interferes with their professional lives. Though many treatments for acne scarring exist including ablative and nonablative lasers, subcision, and peels, none is without risk of adverse effects of pain, post-procedure redness or pigmentary changes. There have been no randomized studies directly comparing the effectiveness and safety profiles of microneedling (Dermapen) to 1,540nm nonablative fractional lasers (Palomar StarLux) in the treatment of atrophic acne scarring in skin of color. This clinical trial aims to determine which treatment modality -- microneedling or nonablative fractional laser -- is safer and more efficacious in the treatment of acne scarring in patients with skin of color.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to dermatology clinic for any reason, or resident or attending dermatologists at Boston University.
* Individuals (men and women) aged 18 and older
* Patients must have atrophic facial acne scarring on the face and desire treatment to improve appearance of acne scarring
* Patients must have Fitzpatrick skin type III-VI
* Patients must be willing to receive five acne scarring treatments at monthly intervals with one follow-up visit to assess for efficacy and adverse effects
* Subjects must speak either English, Chinese, or Spanish.

Exclusion Criteria:

* Subjects who are unable or unwilling to give informed consent.
* Personal history of photosensitivity or photosensitive diseases.
* Pregnancy or breast-feeding.
* Facial surgical or laser treatment in the last 3 months.
* Patients with any active skin infection in the treatment area.
* Coagulopathies or anticoagulant therapy.
* Personal history or presence of hypertrophic scars or keloids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Change in the Goodman and Baron score | Before treatment starts and 3 months after the last/5th treatment
  The Goodman and Baron score considers type of scar, number of scars, and severity of scarring and assigns a grade 1-4 with grade 1 representing mild, macular disease and grade 4 representing severe scarring that is obviously visible at social distances of 50cm, is not easily covered by makeup, and is not able to be flattened by manual stretching of the skin. Lower scores are favorable.

SECONDARY OUTCOMES:
Treatment satisfaction | 3 months after the last/5th treatment
  A questionnaire with questions about participant satisfaction with the treatment, perceived improvement, and perceived adverse effects will be administered at the last visit, 3 months after the treatment is complete. Responses will be compared between the two treatment arms.
Impact of skin disease on the quality of life | 3 months after the last/5th treatment
  Impact of skin disease on the quality of life will be assessed using the Dermatology life Quality Index (DLQI) which is a ten-question questionnaire with responses options of: Very much=3, A lot=2, A little=1, Not at all=0, or Not relevant=0. Range of scores are from 0 to 30 and interpreted as: 0 - 1= no effect at all on patient's life, 2 - 5= small effect on patient's life, 6 - 10= moderate effect on patient's life, 11 - 20= very large effect on patient's life, and 21 - 30= extremely large effect on patient's life. Responses will be compared between the two treatment arms.

CONTACTS AND LOCATIONS:
Overall Officials: Hye Jin Chung, MD, MMS, Principal Investigator — Boston University Department of Dermatology
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No